CLINICAL TRIAL: NCT06970886
Title: Effects of Rhythm-Based Music on Anxiety, Glucose, and Cortisol in Pregnancies With Gestational Diabetes
Brief Title: Effects of Rhythm-Based Music on Pregnancies With Gestational Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esin Ceber Turfan, Professor (Other)
Collaborators: Ege University (Other)
Responsible Party: Sponsor-Investigator, Esin Ceber Turfan, Professor, Dean, Faculty of Health Sciences, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EgeUTYilmaz001
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Anxiety; Blood Sugar; High
Keywords: Anxiety; Blood glucose; Gestational diabetes; Salivary cortisol
MeSH Terms: conditions — Anxiety Disorders; Hyperglycemia; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Since the music intervention in this study will be conducted by the researcher and the cooperation of the pregnant participants is required, masking cannot be applied to the researcher or the participants. To prevent reporting bias during the writing of the research report, masking will be implemented during the statistical analysis and interpretation of the findings. Evaluations will be conducted based on groups labeled as Group I, Group II, and Group III, without revealing the actual group names.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rhythm-Based Active Music Engagement Group (Experimental): Participants will engage in active rhythm-based music making sessions under the guidance of the researcher. Sessions will be conducted once daily for 3 consecutive days. Each session will last approximately 30 minutes and involve creating rhythms using hand drums and body percussion. Participants will follow simple rhythmic patterns designed to promote relaxation and engagement.
  Interventions: Behavioral: Rhythm-Based Music Intervention
- Rhythm-Based Music Listening Group (Experimental): Participants will passively listen to pre-recorded rhythm-based music selected by the researcher. Listening sessions will occur once daily for 3 consecutive days. Each session will last approximately 30 minutes. Participants will be seated comfortably and instructed to focus on the rhythm and flow of the music without actively creating sounds.
  Interventions: Behavioral: Rhythm-Based Music Intervention
- Control Group (No Intervention): Participants in the control group will receive routine prenatal care without any additional music intervention during the study period.

INTERVENTIONS:
Behavioral: Rhythm-Based Music Intervention — The rhythm-based music intervention is designed to reduce anxiety and improve emotional well-being in pregnant women with gestational diabetes. This intervention involves structured music sessions, utilizing rhythm as a therapeutic tool to engage participants in either active creation or passive listening. The intervention aims to promote relaxation, reduce stress, and support overall psychological health by leveraging the emotional and cognitive effects of rhythm and music.
  Arms: Rhythm-Based Active Music Engagement Group; Rhythm-Based Music Listening Group

SUMMARY:
This study is for people who have gestational diabetes, a type of diabetes that happens during pregnancy. People with gestational diabetes may feel more anxious than others during pregnancy. This anxiety can affect their health and their baby's health.

The goal of this study is to see if rhythm-based music can help lower anxiety and improve blood sugar and stress hormone levels. Music may be a safe and low-cost way to support emotional and physical health during pregnancy.

Researchers will test two types of music activities:

Listening to rhythm-based music

Doing rhythm-based music and breathing exercises

The study will include 180 pregnant participants. They will be randomly placed into one of three groups. Each group will be at a different hospital to prevent crossover. Two groups will receive music activities, and the third group will receive usual care.

Participants will stay in the hospital for 3 days. During that time:

Anxiety will be measured on day 1 and day 3 using a short questionnaire

Blood sugar will be measured 3 times a day (morning, afternoon, evening)

Saliva samples will be collected on day 3 to measure cortisol (a stress hormone)

Researchers will also record any medications used by participants.

This study may show that music helps lower anxiety and improve health for people with gestational diabetes. It may also support the use of music as a helpful, non-drug option during pregnancy.

DETAILED DESCRIPTION:
Gestational diabetes is a condition where blood sugar levels become high during pregnancy. This condition can affect both the pregnant person and their baby, leading to health problems during and after pregnancy. People with gestational diabetes often experience higher levels of anxiety. This can make it harder to manage blood sugar and may affect the baby's development.

Music is a safe and low-cost way to support mental and emotional health. Listening to or creating rhythm-based music may help reduce anxiety. Some research shows that music can help people with diabetes, but there are very few studies that look at its effect in pregnancies affected by gestational diabetes.

This study will explore whether rhythm-based music activities can help lower anxiety, blood sugar levels, and cortisol, a hormone related to stress.

A total of 180 pregnant participants with gestational diabetes will be part of the study. They will be randomly assigned to one of three groups:

Group 1: Will listen to rhythm-based music

Group 2: Will take part in guided sessions that include rhythm-based music activities and breathing exercises

Group 3: Will receive standard hospital care without music

Each group will be located at a different hospital in İzmir, Türkiye. This will help prevent participants in different groups from influencing each other.

The music activity will happen over three days, during the participants' hospital stay. Researchers will collect information by:

Measuring anxiety levels using a standard questionnaire on day 1 and day 3

Measuring blood sugar three times a day (morning, afternoon, evening)

Collecting saliva samples to measure cortisol before and after the music activity on day 3

Recording any medications used by participants

This study may show that rhythm-based music is a useful tool to support the health of people with gestational diabetes. If effective, this approach could be used as a non-drug way to lower anxiety and improve health outcomes for both the pregnant person and the baby. The findings could also support using more non-drug, supportive care methods in pregnancy and lead to new research and international collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the study with informed written consent
* Diagnosed with Gestational Diabetes Mellitus (GDM) and currently hospitalised
* In the third trimester of pregnancy
* Over the age of 18
* Have a live, single fetus

Exclusion Criteria:

* Any condition preventing participation in rhythm-based music making and listening (e.g., hearing, vision, or speech impairments)
* Regular and routine music listening habits during pregnancy
* Physical limitations or restrictions
* Mental or cognitive disorders requiring medication
* Use of corticosteroids or medications containing corticosteroids
* Known fetal abnormalities
* Systemic diseases other than GDM (e.g., Hypertension, Type 1 or Type 2 Diabetes, Thyroid disorders, etc.)
* Body mass index (BMI) of 30 or higher
* Discharge from the hospital before the 3rd day of the intervention

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is eligible for female participants only, as it focuses on pregnant women with gestational diabetes.
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-05 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Anxiety Levels | Anxiety levels will be assessed at two time points: Day 1 (Pre-intervention) and Day 3 (Post-intervention). The first measurement will occur before the intervention, and the second will be taken immediately after the 3-day music intervention.
  Anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI), at baseline (Day 1) and post-intervention (Day 3).
  Anxiety level was assessed using the State Anxiety subscale of the State-Trait Anxiety Inventory (STAI-State). The scale consists of 20 items with scores ranging from 20 to 80. Higher scores indicate greater anxiety, representing a worse outcome.

SECONDARY OUTCOMES:
Blood Glucose Levels | Blood glucose levels will be measured three times daily (morning, afternoon, and evening) over the course of 3 consecutive days: Day 1, Day 2, and Day 3. Measurements will be taken at the same time each day to ensure consistency.
  Blood glucose levels will be measured three times per day (morning, afternoon, evening) for 3 consecutive days, using a glucose meter. The average level for each day will be calculated.
Salivary Cortisol Levels | Salivary cortisol levels will be assessed twice on Day 3: once pre-intervention (before the music intervention) and once post-intervention (immediately after the intervention). Saliva samples will be collected at these time points.
  Cortisol levels will be measured twice on Day 3, once before the intervention and once after the intervention, using a salivary cortisol test. Saliva samples will be collected and analyzed to assess changes in cortisol concentration, which serves as an indicator of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Ceber Turfan, Prof, Principal Investigator — Ege University
Locations (1):
- İzmir City Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including outcome measures such as anxiety scores, blood glucose levels, and salivary cortisol levels, will be shared upon reasonable request. Data will be available after publication for qualified researchers conducting academic studies. Access to the data will require approval by the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data will become available 1 year after publication and will be accessible for 5 years.
Access Criteria: Qualified researchers with a sound research proposal and institutional review board (IRB) approval may request access to the de-identified data for academic research purposes. Requests will be evaluated by the principal investigator.

REFERENCES:
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] Adhikari K, Patten SB, Williamson T, Patel AB, Premji S, Tough S, Letourneau N, Giesbrecht G, Metcalfe A. Assessment of anxiety during pregnancy: are existing multiple anxiety scales suitable and comparable in measuring anxiety during pregnancy? J Psychosom Obstet Gynaecol. 2021 Jun;42(2):140-146. doi: 10.1080/0167482X.2020.1725462. Epub 2020 Feb 14. PMID 32056477
- [Background] E Aksoy Y, D Yilmaz S, Kilic S. The effect of music therapy on non-stress test results and anxiety levels in high-risk pregnant women: A randomized controlled trial. Int J Nurs Pract. 2024 Dec;30(6):e13281. doi: 10.1111/ijn.13281. Epub 2024 Jun 20. PMID 39031663
- [Background] Alakidi A, Dimitrov I, Bivolarska AV, Mihaylova V. Changes in the levels of marker molecules salivary alpha-amylase and cortisol as a stress response to everyday activities of general practitioners in rural areas of the Republic of Bulgaria. Rural Remote Health. 2023 Jan;23(1):7318. doi: 10.22605/RRH7318. Epub 2023 Jan 30. PMID 36710477
- [Background] Algül G, Törüner EK. Müzik Temelli Uygulamaların Pediatri Hastalarında Kullanımı ve Hemşirelik Bakımına Etkisi: Geleneksel Derleme. Geleneksel ve Tamamlayıcı Tıp Dergisi.2022; 5(1): 68-74. https://doi.org/10.5336/jtracom.2021-87787
- [Background] Aydemir M, Makaraci Y, Avci B, Urkmez YC, Cintineo HP. The Psychophysiologic Stress and Salivary Cortisol and Alpha-Amylase Awakening Responses to Cross-Country Running Competitions in National-Level Female Athletes. J Strength Cond Res. 2025 May 1;39(5):e676-e683. doi: 10.1519/JSC.0000000000005055. Epub 2025 Mar 4. PMID 40030101
- [Background] Baltaci N, Dogan Yuksekol O, Koc E, Ulucan M. The effects of listening to lullabies and self-selected music at home on prenatal stress and anxiety in nulliparous pregnant women: A randomized-controlled study. Health Care Women Int. 2024;45(5):562-578. doi: 10.1080/07399332.2023.2196510. Epub 2023 Apr 3. PMID 37010820
- [Background] Blair J, Adaway J, Keevil B, Ross R. Salivary cortisol and cortisone in the clinical setting. Curr Opin Endocrinol Diabetes Obes. 2017 Jun;24(3):161-168. doi: 10.1097/MED.0000000000000328. PMID 28375882
- [Background] Castro-Quintas A, Eixarch E, Martin-Gonzalez NS, Daura-Corral M, Marques-Feixa L, Palma-Gudiel H, Rocavert-Barranco M, Miguel-Valero A, Monteserin-Garcia JL, de la Fuente-Tomas L, Crispi F, Arias B, Garcia-Portilla MP, Fananas L. Diurnal cortisol throughout pregnancy and its association with maternal depressive symptoms and birth outcomes. Psychoneuroendocrinology. 2024 Mar;161:106930. doi: 10.1016/j.psyneuen.2023.106930. Epub 2023 Dec 19. PMID 38142606
- [Background] Chang MY, Chen CH, Huang KF. Effects of music therapy on psychological health of women during pregnancy. J Clin Nurs. 2008 Oct;17(19):2580-7. doi: 10.1111/j.1365-2702.2007.02064.x. Epub 2008 Feb 19. PMID 18298503
- [Background] Chang SC, Chen CH. Effects of music therapy on women's physiologic measures, anxiety, and satisfaction during cesarean delivery. Res Nurs Health. 2005 Dec;28(6):453-61. doi: 10.1002/nur.20102. PMID 16287051
- [Background] Correia KF, Dodge LE, Farland LV, Hacker MR, Ginsburg E, Whitcomb BW, Wise LA, Missmer SA. Confounding and effect measure modification in reproductive medicine research. Hum Reprod. 2020 May 1;35(5):1013-1018. doi: 10.1093/humrep/deaa051. PMID 32424412
- [Background] Catalgol S, Ceber Turfan E. The effects of music therapy applied to pregnant women on maternal, fetal, and neonatal results: A randomized controlled study. Health Care Women Int. 2022 May;43(5):448-464. doi: 10.1080/07399332.2021.1944150. Epub 2021 Aug 3. PMID 34344266
- [Background] Devecioğlu F. Müzik Eserlerinde Tempo Terimi ve Metronom Değerlerinin Önemi ve Belirtilmemesinin Oluşturduğu Sorunlar. Akü Amader. 2023; 9(17): 86-143.
- [Background] Dominguez-Solis E, Lima-Serrano M, Lima-Rodriguez JS. Non-pharmacological interventions to reduce anxiety in pregnancy, labour and postpartum: A systematic review. Midwifery. 2021 Nov;102:103126. doi: 10.1016/j.midw.2021.103126. Epub 2021 Aug 14. PMID 34464836
- [Background] Eseadi C, Amedu AN. Potential impact of music interventions in managing diabetic conditions. World J Clin Cases. 2023 May 6;11(13):2916-2924. doi: 10.12998/wjcc.v11.i13.2916. PMID 37215419
- [Background] Estrella-Juarez F, Requena-Mullor M, Garcia-Gonzalez J, Lopez-Villen A, Alarcon-Rodriguez R. Effect of Virtual Reality and Music Therapy on the Physiologic Parameters of Pregnant Women and Fetuses and on Anxiety Levels: A Randomized Controlled Trial. J Midwifery Womens Health. 2023 Jan;68(1):35-43. doi: 10.1111/jmwh.13413. Epub 2022 Nov 16. PMID 36383473
- [Background] Geranmayeh M, Bikdeloo S, Azizi F, Mehran A. Effect of relaxation exercise on fasting blood glucose and blood pressure in gestational diabetes. British Journal of Midwifery. 2019; 27(9): 572-577.
- [Background] Grillo AR, Corneau GM, Vrshek-Schallhorn S. Relationship of cortisol and alpha amylase to behavioral engagement under three levels of negative evaluative psychosocial stress. Psychoneuroendocrinology. 2023 Sep;155:106308. doi: 10.1016/j.psyneuen.2023.106308. Epub 2023 May 30. PMID 37290377
- [Background] Garcia Gonzalez J, Ventura Miranda MI, Requena Mullor M, Parron Carreno T, Alarcon Rodriguez R. Effects of prenatal music stimulation on state/trait anxiety in full-term pregnancy and its influence on childbirth: a randomized controlled trial. J Matern Fetal Neonatal Med. 2018 Apr;31(8):1058-1065. doi: 10.1080/14767058.2017.1306511. Epub 2017 Apr 3. PMID 28287005
- [Background] Gu L, Yang J, Gong Y, Ma Y, Yan S, Huang Y, Wang Y, Peng Y. Lower free thyroid hormone levels are associated with high blood glucose and insulin resistance; these normalize with metabolic improvement of type 2 diabetes. J Diabetes. 2021 Apr;13(4):318-329. doi: 10.1111/1753-0407.13118. Epub 2020 Nov 2. PMID 32981234
- [Background] Gunnar MR, Talge NM, Herrera A. Stressor paradigms in developmental studies: what does and does not work to produce mean increases in salivary cortisol. Psychoneuroendocrinology. 2009 Aug;34(7):953-67. doi: 10.1016/j.psyneuen.2009.02.010. Epub 2009 Mar 24. PMID 19321267
- [Background] Gyasi-Antwi P, Walker L, Moody C, Okyere S, Salt K, Anang L, Eduful E, Laryea D, Ottie-Boakye D, Asah-Opoku K, Asibey S, Sarfo-Kantanka O, Baffour-Agyei E, Shaw I, Adams, G. Global Prevalence of Gestational Diabetes Mellitus: A Systematic Review and Meta-Analysis. New American Journal of Medicine. 2020; 1(3): 1-10.
- [Background] [Hayran O. Bilimsel Araştırmalar Ne Kadar Bilimsel: Karıştırıcılar, Çarpıştırıcılar ve Etki-Ölçüm Değiştiriciler. Journal of Biotechnology and Strategic Health Research. 2021; 5(3): 166-177. https://doi.org/10.34084/bshr.1020533
- [Background] Hinesley J, Cunningham S, Charles R, Olsen K, Masho S, Kornstein S. The Lullaby Project: A Musical Intervention for Pregnant Women. Womens Health Rep (New Rochelle). 2020 Dec 7;1(1):543-549. doi: 10.1089/whr.2020.0084. eCollection 2020. PMID 33786520
- [Background] Hohman EE, Smyth JM, McNitt KM, Pauley AM, Symons Downs D, Savage JS. Urinary cortisol is lower in pregnant women with higher pre-pregnancy BMI. Front Endocrinol (Lausanne). 2023 Jan 11;13:1014574. doi: 10.3389/fendo.2022.1014574. eCollection 2022. PMID 36714602
- [Background] Hussain S. Priya M. Meditation and music intervention for improving pregnancy psychological health. Yoga Mimamsa. 2023; 55(2): 88. https://doi.org/10.4103/ym.ym_34_23
- [Background] Hutchinson JC, Karageorghis CI, Black JD. The Diabeates Project: Perceptual, Affective and Psychophysiological Effects of Music and Music-Video in a Clinical Exercise Setting. Can J Diabetes. 2017 Feb;41(1):90-96. doi: 10.1016/j.jcjd.2016.07.009. Epub 2016 Dec 1. PMID 27916497
- [Background] Ji C, Zhao J, Nie Q, Wang S. The role and outcomes of music therapy during pregnancy: a systematic review of randomized controlled trials. J Psychosom Obstet Gynaecol. 2024 Dec;45(1):2291635. doi: 10.1080/0167482X.2023.2291635. Epub 2023 Dec 26. PMID 38146963
- [Background] Kikkawa M, Shimura A, Nakajima K, Morishita C, Honyashiki M, Tamada Y, Higashi S, Ichiki M, Inoue T, Masuya J. Mediating Effects of Trait Anxiety and State Anxiety on the Effects of Physical Activity on Depressive Symptoms. Int J Environ Res Public Health. 2023 Mar 30;20(7):5319. doi: 10.3390/ijerph20075319. PMID 37047935
- [Background] Kondracki AJ, Valente MJ, Ibrahimou B, Bursac Z. Risk of large for gestational age births at early, full and late term in relation to pre-pregnancy body mass index: Mediation by gestational diabetes status. Paediatr Perinat Epidemiol. 2022 Jul;36(4):566-576. doi: 10.1111/ppe.12809. Epub 2021 Nov 10. PMID 34755381
- [Background] Konsam M, D'Souza SRB, Praharaj SK, Nayak BS, Shetty J, Bhat S, Noronha JA, Panda S. Effectiveness of Music on Perinatal Anxiety Among Pregnant Women and Newborn Behaviors: A Systematic Review and Narrative Synthesis. Indian J Psychol Med. 2023 Nov;45(6):565-572. doi: 10.1177/02537176231167077. Epub 2023 May 6. PMID 38545536
- [Background] Kordi M, Vahed A, Rezaee TF, Mazloum SR, Lotfalizadeh M. Anxiety during Pregnancy and Preeclampsia: A Case-Control Study. Journal of Midwifery and Reproductive Health. 2017; 5(1): 814-820.
- [Background] Lee A, Jang S, Lee S, Park HK, Kim IY, Ahn R, Seok JH, Lee KR. Comparative analysis of salivary cortisol measurements using different assay methods in relation to serum-free cortisol measurement. Pract Lab Med. 2024 Apr 9;40:e00393. doi: 10.1016/j.plabm.2024.e00393. eCollection 2024 May. PMID 38645932
- [Background] Liu YH, Lee CS, Yu CH, Chen CH. Effects of music listening on stress, anxiety, and sleep quality for sleep-disturbed pregnant women. Women Health. 2016;56(3):296-311. doi: 10.1080/03630242.2015.1088116. Epub 2015 Sep 11. PMID 26361642
- [Background] Maul J, Behnam S, Timmesfeld N, Wimberger P. Arabin B. Music during pregnancy: Systematic review to accompany a project to strengthen maternal stress resilience and child outcomes through creative projects. Geburtshilfe und Frauenheilkunde. 2022; 82(10): e123.
- [Background] Mir IA, Chowdhury M, Islam RM, Ling GY, Chowdhury AABM, Hasan ZM, Higashi Y. Relaxing music reduces blood pressure and heart rate among pre-hypertensive young adults: A randomized control trial. J Clin Hypertens (Greenwich). 2021 Feb;23(2):317-322. doi: 10.1111/jch.14126. Epub 2020 Dec 21. PMID 33347732
- [Background] Modzelewski R, Stefanowicz-Rutkowska MM, Matuszewski W, Bandurska-Stankiewicz EM. Gestational Diabetes Mellitus-Recent Literature Review. J Clin Med. 2022 Sep 28;11(19):5736. doi: 10.3390/jcm11195736. PMID 36233604
- [Background] Mumdzic E. Munir A. Perioperative management of diabetes and corticosteroid supplementation. Surgery (Oxford). 2024; 42(4): 266-273.
- [Background] Öner N. LeCompte WA. Durumluk-sürekli kaygı envanteri el kitabı. Boğaziçi Üniversitesi. 1983.
- [Background] Pasternak Y, Miller N, Asali A, Yagur Y, Weitzner O, Nimrodi M, Pasternak Y, Berkovitz A, Biron-Shental T. Does music during labor affect mode of delivery in first labor after epidural anesthesia? A prospective study. Arch Gynecol Obstet. 2019 Nov;300(5):1239-1244. doi: 10.1007/s00404-019-05310-w. Epub 2019 Sep 23. PMID 31549222
- [Background] Pearlmutter P, DeRose G, Samson C, Linehan N, Cen Y, Begdache L, Won D, Koh A. Sweat and saliva cortisol response to stress and nutrition factors. Sci Rep. 2020 Nov 4;10(1):19050. doi: 10.1038/s41598-020-75871-3. PMID 33149196
- [Background] Persico G, Antolini L, Vergani P, Costantini W, Nardi MT, Bellotti L. Maternal singing of lullabies during pregnancy and after birth: Effects on mother-infant bonding and on newborns' behaviour. Concurrent Cohort Study. Women Birth. 2017 Aug;30(4):e214-e220. doi: 10.1016/j.wombi.2017.01.007. Epub 2017 Feb 4. PMID 28169158
- [Background] Qi W, Zhao F, Huang S, Wei Z, Yang H, He K, Li C, Guo Q. Hu J. Effects and Feasibility of a Mindfulness-Based Guqin Music Intervention During Pregnancy on Postpartum Anxiety and Depression: A Pilot Randomized Controlled Trial. Mindfulness. 2023; 14(11): 2641-2656.
- [Background] Qian J, Sun S, Wang M, Sun X, Yu X. Art-based interventions for women's mental health in pregnancy and postpartum: A meta-analysis of randomised controlled trials. Front Psychiatry. 2023 Feb 15;14:1112951. doi: 10.3389/fpsyt.2023.1112951. eCollection 2023. PMID 36873226
- [Background] Qiu C, Sanchez SE, Lam N, Garcia P, Williams MA. Associations of depression and depressive symptoms with preeclampsia: results from a Peruvian case-control study. BMC Womens Health. 2007 Sep 27;7:15. doi: 10.1186/1472-6874-7-15. PMID 17900360
- [Background] Robb SL, Nichols RJ, Ruta RL, Bishop BL. Parker JC. The Effects of Music Assisted Relaxation on Preoperative Anxiety. Journal of Music Therapy. 1995; 32(1): 2-21.
- [Background] Rodrigues KL, Scaranni PODS, Pereira ENGDS, da Silva VVD, Silvares RR, de Araujo BP, Castilho C, Schmidt MI, da Fonseca MJM, Griep RH, Daliry A. Hair cortisol levels are associated with overweight and obesity in the ELSA-Brasil cohort. Front Endocrinol (Lausanne). 2024 Apr 9;15:1361715. doi: 10.3389/fendo.2024.1361715. eCollection 2024. PMID 38654925
- [Background] Salomon R, Weiss S. Relationships Among Number of Stressors, Perceived Stress, and Salivary Cortisol Levels During the Third Trimester of Pregnancy. J Obstet Gynecol Neonatal Nurs. 2024 Mar;53(2):160-171. doi: 10.1016/j.jogn.2023.11.005. Epub 2023 Dec 1. PMID 38048897
- [Background] Sarwar H, Rafiqi SI, Ahmad S, Jinna S, Khan SA, Karim T, Qureshi O, Zahid ZA, Elhai JD, Levine JC, Naqvi SJ, Jaume JC, Imam S. Hyperinsulinemia Associated Depression. Clin Med Insights Endocrinol Diabetes. 2022 Apr 21;15:11795514221090244. doi: 10.1177/11795514221090244. eCollection 2022. PMID 35494421
- [Background] Shahyad S, Rahmani E, Nikdanesh M, Ashoori A, Azadi S. Hassanvandi S. Effectiveness of Neurofeedback on Psychological Stress, Salivary Cortisol and α-amylase Level in Students: A Randomized and Parallel-Group Clinical Trial. Iranian Journal of Psychiatry and Behavioral Sciences. 2024; e140330.
- [Background] Shin HS, Kim JH. Music Therapy on Anxiety, Stress and Maternal-fetal Attachment in Pregnant Women During Transvaginal Ultrasound. Asian Nurs Res (Korean Soc Nurs Sci). 2011 Mar;5(1):19-27. doi: 10.1016/S1976-1317(11)60010-8. Epub 2011 Apr 5. PMID 25029946
- [Background] Soylu N, Bulbul T, Muderris II. The effect of music on fetal well-being and anxiety levels and vital signs of pregnant women during non-stress test: Turkey sample. Health Care Women Int. 2022 May;43(5):499-517. doi: 10.1080/07399332.2021.1973010. Epub 2021 Sep 14. PMID 34520324
- [Background] Spielberger C, Gorsuch R, Lushene R, Vagg P. Jacobs G. Manual for the State-Trait Anxiety Inventory (Form Y1 - Y2). Palo Alto, CA: Consulting Psychologists Press. 1983.
- [Background] Standley JM, Moore RS. Therapeutic effects of music and mother's voice on premature infants. Pediatr Nurs. 1995 Nov-Dec;21(6):509-12, 574. PMID 8700604
- [Background] Stepanek L, Horakova D, Stepanek L, Janout V, Janoutova J, Bouchalova K, Martinik K. Free triiodothyronine/free thyroxine (FT3/FT4) ratio is strongly associated with insulin resistance in euthyroid and hypothyroid adults: a cross-sectional study. Endokrynol Pol. 2021;72(1):8-13. doi: 10.5603/EP.a2020.0066. Epub 2020 Oct 30. PMID 33125689
- [Background] Stoffel M, Neubauer AB, Ditzen B. How to assess and interpret everyday life salivary cortisol measures: A tutorial on practical and statistical considerations. Psychoneuroendocrinology. 2021 Nov;133:105391. doi: 10.1016/j.psyneuen.2021.105391. Epub 2021 Aug 14. PMID 34607270
- [Background] Sunena, Mishra DN. Stress Etiology of Type 2 Diabetes. Curr Diabetes Rev. 2022;18(9):e240222201413. doi: 10.2174/1573399818666220224140934. PMID 35209829
- [Background] Tafet GE, Nemeroff CB. Pharmacological Treatment of Anxiety Disorders: The Role of the HPA Axis. Front Psychiatry. 2020 May 15;11:443. doi: 10.3389/fpsyt.2020.00443. eCollection 2020. PMID 32499732
- [Background] Türkiye Endokrinoloji Ve Metabolizma Derneği (TEMD). Diabetes Mellitus ve Komplikasyonlarının Tanı, Tedavi ve İzlem Kılavuzu (ISBN: 978-625-99759-2-4). 2024.
- [Background] Türkiye Diyabet Vakfı (TDV). Diyabette İnsülin Tedavi Rehberi (ISBN: 978-625-94103-2-6). 2024.
- [Background] Toker E, Komurcu N. Effect of Turkish classical music on prenatal anxiety and satisfaction: A randomized controlled trial in pregnant women with pre-eclampsia. Complement Ther Med. 2017 Feb;30:1-9. doi: 10.1016/j.ctim.2016.11.005. Epub 2016 Nov 18. PMID 28137517
- [Background] Torun Ş. Kanıta Dayalı Müzik Terapisi Uygulamalarında Müziğin Rolü. Anadolu Tıbbı Dergisi. 2022; 1(2): Article 2.
- [Background] van Vliet S, Koh HE, Patterson BW, Yoshino M, LaForest R, Gropler RJ, Klein S, Mittendorfer B. Obesity Is Associated With Increased Basal and Postprandial beta-Cell Insulin Secretion Even in the Absence of Insulin Resistance. Diabetes. 2020 Oct;69(10):2112-2119. doi: 10.2337/db20-0377. Epub 2020 Jul 10. PMID 32651241
- [Background] Vianna P, Bauer ME, Dornfeld D, Chies JA. Distress conditions during pregnancy may lead to pre-eclampsia by increasing cortisol levels and altering lymphocyte sensitivity to glucocorticoids. Med Hypotheses. 2011 Aug;77(2):188-91. doi: 10.1016/j.mehy.2011.04.007. Epub 2011 May 6. PMID 21550175
- [Background] Wang H, Li N, Chivese T, Werfalli M, Sun H, Yuen L, Hoegfeldt CA, Elise Powe C, Immanuel J, Karuranga S, Divakar H, Levitt N, Li C, Simmons D, Yang X; IDF Diabetes Atlas Committee Hyperglycaemia in Pregnancy Special Interest Group. IDF Diabetes Atlas: Estimation of Global and Regional Gestational Diabetes Mellitus Prevalence for 2021 by International Association of Diabetes in Pregnancy Study Group's Criteria. Diabetes Res Clin Pract. 2022 Jan;183:109050. doi: 10.1016/j.diabres.2021.109050. Epub 2021 Dec 6. PMID 34883186
- [Background] Wulff V, Hepp P, Wolf OT, Balan P, Hagenbeck C, Fehm T, Schaal NK. The effects of a music and singing intervention during pregnancy on maternal well-being and mother-infant bonding: a randomised, controlled study. Arch Gynecol Obstet. 2021 Jan;303(1):69-83. doi: 10.1007/s00404-020-05727-8. Epub 2020 Aug 10. PMID 32776296
- [Background] Xie YP, Lin S, Xie BY, Zhao HF. Recent progress in metabolic reprogramming in gestational diabetes mellitus: a review. Front Endocrinol (Lausanne). 2024 Jan 3;14:1284160. doi: 10.3389/fendo.2023.1284160. eCollection 2023. PMID 38234430
- [Background] Yang M, Li L, Zhu H, Alexander IM, Liu S, Zhou W, Ren X. Music therapy to relieve anxiety in pregnant women on bedrest: a randomized, controlled trial. MCN Am J Matern Child Nurs. 2009 Sep-Oct;34(5):316-23. doi: 10.1097/01.NMC.0000360425.52228.95. PMID 19713801
- [Background] Yesilcinar I, Acavut G, Guvenc G. Anxiety during the pregnancy and affecting factors: a cross-sectional study. Arch Gynecol Obstet. 2023 Jan;307(1):301-309. doi: 10.1007/s00404-022-06590-5. Epub 2022 May 18. PMID 35585212
- [Background] Yılmaz B. Can ÜK. Türkiye'de Müzik Terapi Uygulamalarında Kullanılan Müzikler. OPUS International Journal of Society Researches. 2019; 13(19): Article 19.
- [Background] Yılmaz, V. F. Ritim ile Kitle Manipülasyonu. Otuzyedi Sanat ve Tasarım Dergisi. 2022; 1(1): Article 1.
- [Background] Yüksekol ÖD. Başer M. Preeklampsili Gebelerde Kan Basıncının Düzenlenmesi ve Anksiyetenin Azaltılmasında Müziğin Kullanımı. Journal of Academic Research in Nursing. 2021; 7(1): Article 1.
- [Background] Zhao H, Zhang Y, Ye J, Wei H, Huang Z, Ning X, Fu X. A Comparative Study on Insulin Secretion, Insulin Resistance and Thyroid Function in Patients with Polycystic Ovary Syndrome with and without Hashimoto's Thyroiditis. Diabetes Metab Syndr Obes. 2021 Apr 28;14:1817-1821. doi: 10.2147/DMSO.S300015. eCollection 2021. PMID 33953581
- [Background] Zhou LY, Zhang Y, Tian Y, Fu X, Wang LZ, Xie CG. Effect of music intervention on mental health in patients with diabetes mellitus: protocol for a systematic review and meta-analysis of randomizsed controlled trials. BMJ Open. 2020 Aug 20;10(8):e036268. doi: 10.1136/bmjopen-2019-036268. PMID 32819943
- See also: T.C. Strateji ve Bütçe Başkanlığı. "On İkinci Kalkınma Planı (2024-2028)". — http://www.sbb.gov.tr/wp-content/uploads/2023/12/On-Ikinci-Kalkinma-Plani_2024-2028_11122023.pdf
- See also: WHO guide for integration of perinatal mental health in maternal and child health services. — http://www.who.int/publications-detail-redirect/9789240057142
- See also: WHO Traditional Medicine Strategy: 2014-2023. — http://www.who.int/publications-detail-redirect/9789241506096